CLINICAL TRIAL: NCT04222465
Title: Characterizing the Cross-sectional Approach to Investigate the Prevalence of Tissue BRCA1/2 Mutations in Newly Diagnosed Advanced Ovarian Cancer Patients
Acronym: CHRISTELLE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D0817R00018
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Ovarian Neoplasms
Keywords: Advanced ovarian cancer, BRCA1/2
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
This is a multi-center, observational study in Japan. Patients with newly diagnosed FIGO stage III - IV advanced OC will be enrolled sequentially.

In this study, data of 200 subjects will be collected at approximately 20 sites in Japan. To reduce regional bias of study sites, the number of enrolled patients per site will be capped

DETAILED DESCRIPTION:
Study design:This is a multi-center, observational study in Japan. Patients with newly diagnosed FIGO stage III - IV advanced OC will be enrolled sequentially.

In this study, data of 200 subjects will be collected at approximately 20 sites in Japan. To reduce regional bias of study sites, the number of enrolled patients per site will be capped.

Study population:Patients with FIGO stage III - IV epithelial ovarian cancer Drug exposure:Not applicable Planned study sites and sample size:The objective number of patients will be 200 from approximately 20 hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 years or older of Japanese women at the time of consent (the age of death, in case of dead patient)
* Newly diagnosed as advanced OC (FIGO stage III - IV) with epithelial ovarian cancer, primary peritoneal cancer or fallopian-tube cancer [or a combination of these cancers] after January 1, 2019
* Patients who have archived formalin-fixed paraffin-embedded (FFPE) samples of primary or peritoneal metastatic tumor collected after January 1, 2019
* Patients who have undergone or are scheduled to undergo BRACAnalysis
* Patients who give their written informed consent to participate in this study (However, the cases of death should be handled in accordance with the instructions of the Ethical Review Board of each site.)

Exclusion Criteria:

* Patients who are not recommended enrolling this study decided by physician

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Inclusion Criteria: Aged 20 years or older of Japanese women at the time of consent (the age of death, in case of dead patient)
Study Population: This is a Japanese, multi-center, observational study. Patients with newly diagnosed FIGO stage III - IV OC after 1st January, 2019 will be enrolled sequentially.
  Patients those who have undergone or are planning to undergo BRACAnalysis, which detects BRCA mutations, are eligible for this study. In this study, data of 200 subjects will be collected at approximately 20 sites in Japan. To reduce regional bias of study sites, the number of enrolled patients per site will be capped.
Sampling Method: Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

PRIMARY OUTCOMES:
The prevalence of tBRCAm in the newly diagnosed advanced OC patients | Baseline
  For BRCA1 and BRCA2 mutations detected by Myriad myChoice HRD, the number and percentage of patients with the following results will be indicated; deleterious mutation / suspected deleterious / variant of uncertain significance (VUS) / favour polymorphism / no mutation detected

SECONDARY OUTCOMES:
The prevalence of gBRCAm in the subjects | Baseline
  For BRCA1 and BRCA2 mutations detected by BRACAnalysis, the number and percentage of patients with the following results will be indicated; deleterious mutation / suspected deleterious / variant of uncertain significance (VUS) / favour polymorphism / no mutation detected
The prevalence of sBRCAm in the subjects | Baseline
  For BRCA1 and BRCA2 mutations detected by BRACAnalysis and Myriad myChoice HRD, the number and percentage of patients with the following results will be indicated; deleterious mutation / suspected deleterious
The ratio of sBRCAm out of tBRCAm | Baseline
  Calculate the rate of sBRCAm out of tBRCAm

OTHER OUTCOMES:
tBRCA variant description | Baseline
  BRCA1 and BRCA2 variants detected by Myriad myChoice HRD (location and type of mutation) will be described.

CONTACTS AND LOCATIONS:
Locations (20):
- Japan (20):
  - Research Site, Matsuyama, Ehime
  - Research Site, Tōon, Ehime
  - Research Site, Yoshida, Fukui
  - Research Site, Kitakyushu, Fukuoka
  - Research Site, Sapporo, Hokkaido
  - Research Site, Amagasaki, Hyōgo
  - Research Site, Kobe, Hyōgo
  - Research Site, Tsukuba, Ibaraki
  - Research Site, Sendai, Miyagi
  - Research Site, Kashihara, Nara
  - Research Site, Izumo, Shimane
  - Research Site, Bunkyo, Tokyo
  - Research Site, Minato, Tokyo
  - Research Site, Musashino, Tokyo
  - Research Site, Shinjuku, Tokyo
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Kumamoto
  - Research Site, Niigata
  - Research Site, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials/studies via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0817R00018&attachmentIdentifier=a30ddc24-73b1-4b02-9d54-a405bf03ff2d&fileName=D0817R00018_CHRISTELLE_CSRsynopsis.pdf&versionIdentifier=